CLINICAL TRIAL: NCT01504568
Title: The Use of Prophylactic Antibiotics in Isolated Blowout Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 134357
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Orbital Fractures; Orbital Cellulitis
MeSH Terms: conditions — Orbital Fractures; Orbital Cellulitis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic Antibotics (Other): Amoxicillin/clavulanic acid
  Interventions: Other: Treatment
- Non Treatment (No Intervention): Subjects will be followed without the use of antibiotics.

INTERVENTIONS:
Other: Treatment — Adults: ≥40 kg:250mg every eight hours Children: <40kg: 20mg/kg/day divided in three doses (up to 250mg) every eight hours Suspension form 250mg/ml
  Other Names: Amoxcillin/cavulanic acid
  Arms: Prophylactic Antibotics

SUMMARY:
The purpose of the research is to perform a quality assurance evaluation using randomized prospective analysis the rate of orbital cellulitis as a complication of nonsurgical orbital blowout fracture in patients treated versus not treated with prophylactic antibiotics.

The investigators goal is to show the use of prophylactic antibiotics in orbital blowout fractures does not significantly decrease the rate of orbital cellulitis and is thus not indicated.

DETAILED DESCRIPTION:
Orbital fractures are a common occurrence in association with a wide variety of blunt trauma injuries to the face. One type of fracture is that involving the orbital floor, or an isolated blowout fracture. One common current practice is to use prophylactic antibiotics in these cases to prevent the theoretical occurrence of an orbital cellulitis originating from sinus flora, though there is no current standard of care regarding this practice. Many surgeons may elect to not use antibiotics for this very reason.

The use of prophylactic antibiotics in isolated blowout fractures where there is no occlusion of the ostium is not defined, and no prospective controlled study has been undertaken to suggest the most appropriate course of action to take. Our goal in this study is to determine a correct course of action for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Isolated orbital blow out fracture in patients between the ages 5 to 99 years old

Exclusion Criteria:

* Involvement of the orbital rim in the floor fracture requiring the use of antibiotics
* Involvement of the orbital rim in the floor fracture
* Radiographic evidence of occlusion of the maxillary sinus ostium
* Determined need for surgical intervention or prior use of synthetic implanted material in or around the involved maxillary sinus
* Any symptoms of sinonasal disease in the preceding 3 month for any reason
* Any use of oral or IV antibiotics in the preceding 3 month for any reason
* Documented allergy to penicillin or amoxicillin prohibiting its use
* Any currently immunosuppressed state, including actively treated autoimmune disease; use of steroids, immunomodulatory medication, or chemotherapy within the last year; diagnosis of active cancer within the last year

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Orbital Cellulitis | Two weeks
  The rate of orbital cellulitis as a complication of nonsurgical orbital blowout fracture in patients treated versus not treated with prophylactic antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Westfall, M.D., Principal Investigator — University of Arkansas; Bradley Thuro, M.D., Principal Investigator — University of Arkansas; John Pemberton, D.O., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States